CLINICAL TRIAL: NCT02582268
Title: Introducing Trans- Abdominal Guided Intrauterine Device Insertion, a Single Blinded Randomized Control Trial
Brief Title: A Novel IUD Insertion Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Lecturer of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CU151020
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAS guided IUD insertion (Experimental): the female will be asked to be full bladder. the trans-abdominal probe will be placed by an assistant on the suprapubic region. under speculum examination, the intrauterine device IUD (TCu 380A) will be placed till it reaches the fundus of the uterus and then released.
  Interventions: Device: intrauterine device TCu 380A; Radiation: Trans-abdominal sonography
- Traditional IUD insertion (Experimental): the intrauterine device TCu 380A will be inserted in the conventional method, and checked afterwards by transvaginal ultrasound. the trans-abdominal probe will also be placed by an assistant on the suprapubic region ( the image would be on freeze mode) as it is not actually used , it is just to make the same settings for the participant females.
  Interventions: Device: intrauterine device TCu 380A

INTERVENTIONS:
Device: intrauterine device TCu 380A
  Other Names: TCu 380A
Radiation: Trans-abdominal sonography
  Other Names: TAS
  Arms: TAS guided IUD insertion

SUMMARY:
A previous trial performed by our research team, in order to reduce the pain associated with intrauterine device insertion, compared the novel technique of IUD insertion under the guidance of the trans-abdominal sonography to the traditional method of IUD insertion. It came up with the conclusion that the TAS guided IUD insertion is significantly lower in pain score and time taken for insertion, when compared with the traditional method. In this study our researchers aim to abolish the distracting effect of the technician and the TAS probe (which might have interfered with previous results).

ELIGIBILITY:
Inclusion Criteria:

* Females desiring contraception with the use of IUD
* Females with history of previous vaginal delivery

Exclusion Criteria:

* Are pregnant or think they may be pregnant
* Septic pregnancy or abortion
* Have unexplained abnormal vaginal bleeding
* Have untreated cervical cancer
* Have malignant gestational trophoblastic disease
* Have uterine cancer
* Have uterine abnormalities
* Have or may have had a pelvic infection within the past three months
* Have or may have any sexually transmitted disease
* Have pelvic tuberculosis
* Are postpartum between 48 hours and 4 weeks
* Have benign gestational trophoblastic disease

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
degree of pain during IUD insertion | 4 months
  Pain will be assessed by the use of visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Dakhly DMR, Bassiouny YA. Ultrasound-guided intrauterine device insertion: a step closer to painless insertion: a randomized control trial. Eur J Contracept Reprod Health Care. 2017 Oct;22(5):349-353. doi: 10.1080/13625187.2017.1381234. Epub 2017 Oct 5. PMID 28978240